CLINICAL TRIAL: NCT03260725
Title: Evaluating the Feasibility of Internet-delivered Parent-Child Interaction Therapy
Brief Title: Evaluating the Feasibility of Internet-delivered PCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-13-0451-CR01
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder; Disruptive Behavior Disorder Nos
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Intervention Model Description: Internet-delivered treatment v. clinic-delivered treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered treatment (Experimental): This treatment arm entails Internet-Delivered PCIT (I-PCIT) remotely delivered in real time using videoconferencing. Families stream live parent-child interactions from their own home to a remote therapist who provides live bug-in-the-ear parent coaching via a parent-worn Bluetooth earpiece.
  Interventions: Behavioral: Internet-delivered PCIT (I-PCIT)
- Clinic-delivered treatment (Active Comparator): This treatment arm entails Parent-Child Interaction Therapy (PCIT) delivered in the clinic. For much of the treatment, the therapist observes family interactions from behind a 1-way mirror and provides live bug-in-the-ear parent coaching via a parent-worn earpiece.
  Interventions: Behavioral: Parent-Child Interaction Therapy (PCIT)

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy (PCIT) — PCIT is a short-term intervention that incorporates principles of play therapy into behavioral parent training, drawing on attachment and social learning theories to emphasize positive attention, consistency, problem solving, and communication. Treatment is delivered in the clinic.
  Arms: Clinic-delivered treatment
Behavioral: Internet-delivered PCIT (I-PCIT) — I-PCIT is a short-term intervention that incorporates principles of play therapy into behavioral parent training, drawing on attachment and social learning theories to emphasize positive attention, consistency, problem solving, and communication. Treatment is delivered to families in their own home in real-time via videoconferencing over the Internet by a remote therapist.
  Arms: Internet-delivered treatment

SUMMARY:
The present study is leveraging a randomized-controlled design to evaluate an Internet-based format for the delivery of Parent-Child Interaction Therapy (I-PCIT). Drawing on videoteleconferencing technology, this format affords real-time interactions for the provision of care traditionally delivered in person, regardless of a family's geographic proximity to a mental health facility. Moreover, drawing on technological innovation to deliver interventions directly to families in their natural settings may extend the ecological validity of PCIT, as treatment is delivered in the very context in which child problems occur. Families seeking treatment for early child disruptive behavior problems (N=40) are being randomly assigned to either receive Internet-delivered PCIT or clinic-based PCIT. Outcomes and feasibility/acceptability will be assessed across the treatment phase as well as at post-treatment and 6-month follow-up.

DETAILED DESCRIPTION:
Establishing the feasibility of an Internet-based format for the delivery of evidence-based parent management is a critical step in the evaluation of technological innovations and their potential for advancing children's mental health care. Drawing on teleconferencing technology, such a format affords real-time interactions for the provision of care traditionally delivered in person, regardless of a family's geographic proximity to a mental health facility. Moreover, drawing on technological innovation to deliver interventions directly to families in their natural settings may extend the ecological validity of treatments, as treatments are delivered in the very contexts in which child problems occur.

The objective of the present study is to develop an Internet-delivered Parent-Child Interaction Therapy (PCIT) protocol for preschoolers with Oppositional Defiant Disorder (ODD) or Conduct Disorder (CD) and to evaluate via randomized controlled trial (RCT) the feasibility and acceptability of enrolling, retaining, and treating children with I-PCIT relative to traditional PCIT. Phase I will involve development of an Internet-delivered PCIT (I-PCIT) protocol and treatment materials, including therapist treatment manual and online session handouts. Phase II will entail a case series: the PI will treat 5 consecutive preschool ODD/CD cases with I-PCIT, affording opportunity to further work out any difficulties with protocol or equipment. Phase III will entail testing the feasibility and acceptability of I-PCIT in a pilot RCT conducted with 40 children (ages 3-5) meeting for a Diagnostic and Statistical Manual (DSM-IV) principal diagnosis of ODD or CD and their parent(s) randomly assigned to I-PCIT or traditional PCIT. Parents will provide informed consent. All eligible families will receive evidence based treatment. Treatment will either be either in-clinic Parent-Child Interaction Therapy (PCIT) or Internet-delivered PCIT (I-PCIT). Formal evaluations will be conducted at baseline, post-treatment, and 6-month follow-up. Families can opt to participate in two optional psychophysiological components of the study (one involving behavioral tasks while parents are monitored via physiological equipment, and one involving play tasks while children are monitored via physiological equipment). All assessments will be conducted in the Department of Psychology at Florida International University (FIU), in the Center for Children and Families.

ELIGIBILITY:
Inclusion Criteria:

* Children (ages 3-5) meeting for DSM-IV principal Oppositional Defiant Disorder (ODD) or Conduct Disorder (CD), and at least 1 primary caretaker.
* Eyberg Child Behavior Inventory-Intensity Score in clinical range (i.e., >132).
* English-speaking (child & caretakers).
* Family home equipped w/ broadband connection and computer equipped with Pentium (or compatible) processor, 128 MB random-access memory (RAM), 200 Megabytes available of hard disk space, 16-bit color display adapter, universal series bus (USB) port.

Exclusion Criteria:

* Behavior problems due to organic pathology or trauma,
* Child receiving medication to manage behavior difficulties,
* Presence of child emotional/behavior problem more impairing than ODD or CD,
* Parent or child score <75 standard score on intelligence quotient (IQ) screening,
* History of severe physical or mental impairments (e.g., mental retardation, deafness, blindness, pervasive developmental disorder) in child or participating caretaker(s).
* Child is a ward of the state

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions (CGI) Improvement Scale | Post-treatment (average = 35.2 weeks)
  Most widely used clinician-rated measure of treatment-related changes in functioning. The CGI-Improvement rates improvement on a 7-point scale, ranging from 1 ("very much improved") to 7 ("very much worse"). CGI-Improvement scores of 1 ("very much improved") or 2 ("much improved") reflect "treatment response." CGI-Improvement scores of 1 ("very much improved") reflect "excellent response." Completed by Independent Evaluator (IE) in present study.

SECONDARY OUTCOMES:
Eyberg Child Behavior Inventory (ECBI) | Baseline, post treatment (average = 35.2 weeks), and 6 month follow-up
  Parent-report of child behavior problems that yields an Intensity Score (indicating frequency of symptoms, scores over 132 reflect clinical range) and Problem Score (indicating how problematic symptoms are for caregivers).
Kiddie Disruptive Behavior Disorders Schedule (K-DBDS) | Baseline, post treatment (average = 35.2 weeks), and 6 month follow-up
  A supported parent interview that covers ODD, CD, and Attention-Deficit/Hyperactivity Disorder (ADHD), in preschoolers.
  Items are worded to maximize DSM-IV consistency, while retaining developmental appropriateness.
Barriers to Treatment Participation Scale (BTPS) | Mid-treatment (average = 17.2 weeks) and post treatment (average = 35.2 weeks)
  44-item parent-report measure of perceived barriers to treatment participation. Items are rated along 5-point scales and assess stressors and obstacles that compete with treatment (e.g., transportation, scheduling), treatment demands issues (e.g., uncomfortable treatment setting), and attitudes about treatment and the therapist (e.g., treatment is not working). Tallying the items yields a total barriers score
Children's Global Assessment Scale (CGAS) | Baseline, post-treatment (average = 35.2 weeks), and 6 month follow-up
  Clinician-rated index of functioning. Scores range from 0-100; lower scores indicate greater impairment.
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (average = 35.2 weeks)
  Assessment of consumer satisfaction with services. Used as a parent report in present study
Therapy Attitude Inventory (TAI) | Posttreatment (average = 35.2 weeks)
  Parent-report of satisfaction with parent training
Child Behavior Checklist for ages 1.5 to 5 (CBCL 1.5-5) | Baseline, mid-treatment (average = 17.2 weeks), post treatment (average = 35.2 weeks), and 6 month follow-up
  Standardized instrument for assessing behavioral and emotional problems in young children, demonstrating very strong psychometric properties. Empirically based scales, normed for age and sex, are generated. T-scores below 65 reflect normative functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will use a controlled access approach, using a robust system to review requests and provide secure access to de-identified data.